CLINICAL TRIAL: NCT03387631
Title: Efficacy and Safety of Artemether Lumefantrine for the Treatment of Uncomplicated Malaria in Tanzania
Brief Title: Efficacy And Safety Of AL For The Treatment Of Uncomplicated Falciparum Malaria In Mainland Tanzania
Acronym: TES2016
Status: Completed | Type: Observational
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Dr. Celine Mandara, Research Sientist, National Institute for Medical Research, Tanzania
Other Study IDs: NIMRTanzania
Record Dates: First submitted 2017-02-21; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-02

CONDITIONS: Uncomplicated Malaria
Keywords: Efficacy safety uncomplicated malaria AL
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Artemether-Lumefantrine
  Other Names: Coartem

SUMMARY:
Following the development of drug resistance to antimalarial first line treatment of uncomplicated malaria with SP by P.falciparum in mainland Tanzania, the Ministry of Health - Tanzania, introduced ACTs with AL as first line treatment for uncomplicated falciparum malaria in 2006. In the advent of wide scale deployment of ACT together with strengthened vector control with LLIN in mainland Tanzania, there is a trend of shrinking the burden of malaria. The decline of outpatient malaria cases in recent years and declining entomological inoculation rates (EIR) that are currently being recorded in most areas that were before considered to be holo/hyper-endemic to malaria transmission is another indicator of the shift in the epidemiology of malaria transmission in Tanzania. This current shift provides a new and yet critical challenge with regards to assessment and monitoring of the efficacy of the first-line treatment specifically considering that artemisinin resistance has been confirmed in the Greater Mekong sub-region. The aim of the study was to set up a system for country wide representative surveillance to obtain data of the safety and efficacy of AL following countrywide use of ACTs for treatment of uncomplicated malaria in Tanzania. The study was conducted in the framework of the existing NMCP sentinel sites that are ecological representative for malaria endemicity in Tanzania Objective: To assess the efficacy and safety of artemether-lumefantrine, artesunate-amodiaquine and dihydroartemisinin-piperaquine for the treatment of uncomplicated falciparum malaria in Tanzania.

Methods: The study was conducted in eight sentinel sites of NMCP (Kyela, Mkuzi, Kibaha, Ujiji, Nagaga, Chamwino, Igombe and Mlimba) in mainland Tanzania. Four sentinel sites (Mlimba, Mkuzi, Kibaha, and Ujiji) were covered in 2016 and the rest will be involved in the second round to be undertaken in 2017.

Patients were treated with AL for 3 days and the study was conducted from April to Sept 2016. The results of this study will assist the Ministry of Health to monitor the efficacy and safety of the ACTs in Tanzania, provide baseline data on parasite clearance time and for assessing the current national treatment guidelines for uncomplicated falciparum malaria.

DETAILED DESCRIPTION:
The study was on safety and efficacy of artemether lumefantrine for the treatment of uncomplicated malaria, to be done in 8 National Malaria Control Programme sentinel sites The study was proposed to be done in 2 phases; the first phase in Mkuzi, Ujiji, Kibaha and Mlimba fro April 2016-Sept 2016 The second phase to be done in the other 4 sites of Igombe, Chwamwino, Kyela and Nagaga from February - October 2017

ELIGIBILITY:
Inclusion Criteria: • Patients aged 6 months-10 years.

* mono-infection with P. falciparum detected by microscopy;
* parasitaemia of 250 - 200,000/μl asexual forms;
* presence of axillary temperature ≥37.5 °C or history of fever during the past 24 hours
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the parents or guardians of children.

Exclusion Criteria:

* presence of general danger signs in children aged 6 months-10 years or signs of severe falciparum malaria according to the definitions of WHO (Appendix 1);
* weight under 5 Kg
* mixed or mono-infection with another Plasmodium species detected by microscopy;
* presence of severe malnutrition (defined as a child who has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm);
* presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* regular medication, which may interfere with antimalarial pharmacokinetics;
* history of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients aged 6 months-10 years and with uncomplicated falciparum malaria presenting at the study health clinics. Parents or guardians will give informed consent on behalf of their children.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cure rates as per WHO protocol | 28 days
  number with ACPR

CONTACTS AND LOCATIONS:
Overall Officials: Deusdedith S Ishengoma, PhD, Principal Investigator — National Institute for Medical Research

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ishengoma DS, Mandara CI, Francis F, Talundzic E, Lucchi NW, Ngasala B, Kabanywanyi AM, Mahende MK, Kamugisha E, Kavishe RA, Muro F, Mohamed A, Mandike R, Mkude S, Chacky F, Paxton L, Greer G, Kitojo CA, Njau R, Martin T, Venkatesan M, Warsame M, Halsey ES, Udhayakumar V. Efficacy and safety of artemether-lumefantrine for the treatment of uncomplicated malaria and prevalence of Pfk13 and Pfmdr1 polymorphisms after a decade of using artemisinin-based combination therapy in mainland Tanzania. Malar J. 2019 Mar 21;18(1):88. doi: 10.1186/s12936-019-2730-1. PMID 30898164